CLINICAL TRIAL: NCT03356275
Title: Mobile Coach for Parents of Children and Adolescents With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: BodiMojo, Inc. (Other)
Responsible Party: Principal Investigator, Lonnie Zeltzer, Distinguished Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: R43HD090774 (NIH)
Record Dates: First submitted 2017-11-21; First posted 2017-11-29 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Parents; Chronic Pain; Pediatric Disorder
MeSH Terms: conditions — Chronic Pain | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobile application (Experimental): Psychosocial support for parents, including: brief audio mindfulness recordings, videos, and psychoeducational materials.
  Interventions: Behavioral: Mindfulness for Resilience in Illness: Support for Parents

INTERVENTIONS:
Behavioral: Mindfulness for Resilience in Illness: Support for Parents — Mobile application focusing on emotional coping skills for parents of children and adolescents with chronic pain. Components of the module include: library of mindfulness meditations/relaxations; peer support videos; and psychoeducational information related to pain, stress, and mindfulness.

SUMMARY:
Chronic pain is estimated to affect 20% to 35% of children and adolescents around the world, and is associated with increased risk of anxiety and depression among children and adolescents, as well as coping challenges, anxiety, depression, and anger in their parents. For parents, learning to manage stress is critical, as parents play a significant role in a child's experience of pain. Parental behaviors such as over-involvement, solicitousness and rejection are associated with decreased functioning, including higher school absenteeism in children and teens. A number of interventions demonstrate that teaching skills to parents can have a direct and positive impact on the health of children and adolescents with chronic pain. The investigators propose to create and test the BodiMojo Parent Buddy which will provide parents with real-time, tailored and adaptive coping and stress management support and will provide a curriculum of skills for responding to a child in pain in order to promote child functioning.

Thirty parents of children ages 8-18 who have been diagnosed with a non-cancer chronic pain condition will participate in this user-testing study. Parents will complete a brief set of questionnaires before and after the intervention, and will be instructed to open and use the app each day for 30 days. Participants will complete audio mindfulness exercises, watch brief video clips, and read psychoeducational information about pain, coping, and communication skills. Post-intervention questionnaires will also include an acceptance test to assess participants' opinions about the helpfulness and usability of the app. Parent participation is expected to take around 3.5 hours total over the 30 day study period.

ELIGIBILITY:
Inclusion Criteria:

* Parents who self-report parenting a child or adolescent ages 8-18 with non-cancer chronic pain.
* Daily use of a smartphone (iOS, Android, or Windows) or tablet.
* Ability to speak and understand English.

Exclusion Criteria:

* Inability to provide consent
* Inability to speak and understand English

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2018-03-13 (Actual); Study Completion 2018-03-13 (Actual)

PRIMARY OUTCOMES:
Ratio of the days during the 30-day intervention period during which participants use the app | At the conclusion of the final day of the intervention (Day 30)
  Determined by how often participants engaged and used certain features. To be considered feasible, participants must have opened the app on at least half of the days.
Acceptance | Within 7 days of competing the intervention
  Determined by participants' responses to acceptance test questions in the following domains: (1) how much the participant liked the various app features; (2) how much participants liked the video and supplementary content; and (3) helpfulness of various app features. Responses will be given on a one to seven-point-scale ranging "terrible" to "excellent." The intervention will be deemed acceptable if at least 80% of participants rate each question an average of at least "5" ("good") on the 7-point scale.

CONTACTS AND LOCATIONS:
Overall Officials: Lonnie K Zeltzer, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Pediatric Pain and Palliative Care Program Research Offices, Los Angeles, California, United States